CLINICAL TRIAL: NCT01188252
Title: An Open-label, Phase I, Dose-escalation Study to Characterize the Safety, Tolerability, Pharmacokinetics, and Maximum Tolerated Dose of BAY 1000394 Given Twice Daily in a 3 Days on / 4 Days Off Schedule in Subjects With Advanced Malignancies
Brief Title: Clinical Study to Evaluate the Maximum Tolerated Dose of BAY1000394 Given in a 3 Days on / 4 Days Off Schedule in Subjects With Advanced Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14484; 2010-019191-79 (EudraCT Number)
Record Dates: First submitted 2010-07-30; First posted 2010-08-25 (Estimated); Last update posted 2017-01-09 (Estimated); Status verified 2017-01

CONDITIONS: Neoplasms
Keywords: Phase I; Dose escalation; Kinase inhibitor; Cyclin-dependent kinases
MeSH Terms: conditions — Neoplasms | interventions — roniciclib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Roniciclib (Experimental)
  Interventions: Drug: Roniciclib (BAY1000394)

INTERVENTIONS:
Drug: Roniciclib (BAY1000394) — Oral administration twice daily in a 3 days on / 4 days off schedule. Starting dose will be 0.3 mg corresponding to approximately 0.005 mg/kg and dose will be escalated dependent on any dose limiting toxicities.

SUMMARY:
Clinical study to determine safety, tolerability, to measure how the drug is metabolized by the body and to determine the maximum tolerated dose of BAY1000394 given in an intermittent 3 days on / 4 days off schedule to patients with advanced malignancies

ELIGIBILITY:
Inclusion Criteria:

* Eastern Cooperative Oncology Group (ECOG) performance status of 0 - 1
* Life expectancy of at least 12 weeks
* Subjects with advanced, histologically or cytologically confirmed solid tumors, refractory to any standard therapy, have no standard therapy available, or subjects must have actively refused any treatment which would be regarded standard, and / or if in the judgment of the investigator, experimental treatment is clinically and ethically acceptable
* At least 1 tumor lesion measurable by computer tomography (CT) scan or magnetic resonance imaging (MRI) according to RECIST 1.1
* Adequate bone marrow, liver, and renal functions as assessed by the following laboratory requirements to be conducted within 14 days prior to the first dose of study drug

Exclusion Criteria:

* History of cardiac disease: congestive heart failure > NYHA Class II, unstable angina (anginal symptoms at rest), any episodes of angina or history of myocardial infarction, cardiac arrhythmias requiring anti-arrhythmic therapy (beta blockers or digoxin are permitted), previous venous or arterial thrombotic events, pulmonary embolism
* Moderate or severe hepatic impairment, i.e. Child-Pugh class B or C(3)
* History of human immunodeficiency virus (HIV) infection or chronic hepatitis B or C
* Active clinically serious infections of CTCAE > Grade 2 (CTCAE v4.02)
* Symptomatic metastatic brain or meningeal tumors unless the subject is > 3 months from definitive therapy, has no evidence of tumor growth on an imaging study within 4 weeks prior to study entry, and is clinically stable with respect to the tumor at the time of study entry. Subjects must not be on acute steroid therapy or taper off steroid therapy (chronic steroid therapy is acceptable provided that the dose is stable for 4 weeks prior to study entry and following screening CT / MRI scan). Subjects with neurological symptoms should undergo a CT / MRI scan of the brain to exclude new or progressive brain metastases. Spinal cord metastasis is acceptable
* Seizure disorder requiring therapy (such as steroids or anti-epileptics)
* History of organ allograft
* Evidence or history of bleeding disorder, i.e. any hemorrhage / bleeding event of CTCAE > Grade 2 within 4 weeks prior to prior to the first dose of study drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2010-08; Primary Completion 2016-06 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Safety: Frequency of adverse events | Up to 3 years or longer if indicated
Maximum tolerated dose: Measured by adverse event profile | Up to 3 years or longer if indicated
Pharmacokinetics: Plasma concentrations of BAY1000394 will be measured. The following parameters will be calculated: Cmax, tmax, AUC(0-tn), AUC, and half-life. | Approximately 6 weeks

SECONDARY OUTCOMES:
Biomarkers evaluation: analysis of apoptosis marker CK18/M30 and total soluble cytokeratin CK18/M65 | Up to 3 years or longer if indicated
Assessment of expression (IHC) and amplification status (FISH) of markers related to cell proliferation and the cell cycle in Paraffin-embedded archival tumor samples. These will include, but may not be limited to Cyclin E, Cyclin D, p21, and Ki67 | From archival tumor blocks
Functional testing of peripheral leucocytes, for example induction of cytokine synthesis | Approximately 6 weeks
Assessment of intracellular biomarkers of apoptosis (for example activated caspase 3, annexin V, expression of MCL 1 for patients with chronic lymphocytic leucemia only | Approximately 6 weeks
Tumor response evaluation based on RECIST 1.1 (solid tumors) or response based on the pertinent guidelines (malignant lymphoma, chronic lymphocytic leukemia) every 2 cycles | Up to 3 years or longer if indicated

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (9):
- United States (3):
  - St Louis, Missouri
  - Buffalo, New York
  - Cleveland, Ohio
- France (4):
  - Caen
  - Lyon
  - Marseille
  - Villejuif
- Germany (2):
  - Heidelberg, Baden-Wurttemberg
  - Herne, North Rhine-Westphalia